CLINICAL TRIAL: NCT01008410
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Assess the Efficacy and Safety of Budesonide Foam (2 mg/25 mL BID for 2 Weeks, Followed by 2 mg/25 mL QD for 4 Weeks) Versus Placebo in Subjects With Active Mild to Moderate Ulcerative Proctitis or Proctosigmoiditis
Brief Title: Efficacy and Safety of Budesonide Foam for Participants With Active Mild to Moderate Ulcerative Proctitis or Proctosigmoiditis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BUCF3001
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Proctitis; Proctosigmoiditis
Keywords: Proctitis; Proctosigmoiditis; Ulcerative; Salix; Budesonide foam; Budesonide; Rectal; Gastrointestinal; Colitis; UC; UP; UPS; Additional relevant MeSH terms:; Proctocolitis; Ulcer; Colitis, Ulcerative; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Rectal Diseases; Intestinal Diseases; Colonic Diseases; Sigmoid Diseases; Pathologic Processes; Inflammatory Bowel Diseases; Bronchodilator Agents; Autonomic Agents; Peripheral Nervous System Agents; Physiological Effects of Drugs; Pharmacologic Actions; Anti-Asthmatic Agents; Respiratory System Agents; Therapeutic Uses; Glucocorticoids; Hormones; Hormones, Hormone Substitutes, and Hormone Antagonists; Anti-Inflammatory Agents
MeSH Terms: conditions — Proctitis; Proctocolitis; Ulcer; Colitis; Colitis, Ulcerative; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Rectal Diseases; Intestinal Diseases; Colonic Diseases; Sigmoid Diseases; Pathologic Processes; Inflammatory Bowel Diseases | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Budesonide (Experimental): Participants who were diagnosed with active mild to moderate UP or UPS, will receive 2 milligrams (mg)/25 milliliter (mL) of budesonide foam, rectally twice daily for a period of 2 weeks followed by 2 mg/25 mL of budesonide foam, rectally once daily for a period of 4 weeks.
  Interventions: Drug: Budesonide
- Placebo (Placebo Comparator): Participants who were diagnosed with active mild to moderate UP or UPS will receive 25 mL of placebo matching to budesonide foam twice daily for a period of 2 weeks followed by once daily for a period of 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide — Budesonide will be administered as per the dose and schedule specified in the respective arm.
  Arms: Budesonide
Drug: Placebo — Placebo matching to budesonide will be administered as per the schedule specified in the respective arm.
  Arms: Placebo

SUMMARY:
The purpose of this study is to establish the efficacy profile of rectally administered budesonide foam, as compared to an equivalent volume of rectally administered placebo foam over the same dosing schedule, in participants who present with a diagnosis of active, mild to moderate, ulcerative proctitis (UP) or ulcerative proctosigmoiditis (UPS). During the study, eligible participants will be allowed to maintain previously established oral 5-aminosalicylic acid (5-ASA) treatment at doses up to 4.8 grams/day (g/day).

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign written informed consent.
* Male or non-pregnant and non-lactating females.
* Confirmed diagnosis (by endoscopy procedure) of active, mild to moderate UP or UPS, with disease extending at least 5 centimeters (cm) but no further than 40 cm from the anal verge.
* Must possess a baseline Modified Mayo Disease Activity Index (MMDAI) score between 5 and 10.

Exclusion Criteria:

* History or current diagnosis of Crohn's disease and indeterminate colitis.
* Prior gastrointestinal surgery except appendectomy and hernia.
* Concomitant active gastrointestinal disease or distortion of intestinal anatomy.
* History of diverticulitis, collagenous colitis, celiac disease, recurrent pancreatic or known gallbladder disease.
* Uncontrolled, previously diagnosed type 1 or 2 diabetes mellitus.
* Uncontrolled abnormal thyroid function.
* Unstable significant cardiovascular, endocrine, neurologic or pulmonary disease.
* Hemoglobin levels less than (<) 7.5 grams /deciliter (g/dL).
* History of sclerosing cholangitis, cirrhosis, or hepatic impairment.
* Renal disease manifested by greater than (>) 2.0 milligrams/deciliter (mg/dL) serum creatinine.
* History of avascular hip necrosis, active tuberculosis, ocular herpes simplex or ocular varicella zoster, malignant disease, and human immunodeficiency virus (HIV) or hepatitis B or C.
* Adrenal insufficiency.
* Active systemic or cutaneous infection or toxic megacolon, fistula, perforation or abscess.
* History of uncontrolled psychiatric disorders or seizure disorders.
* History of asthma requiring ongoing use of inhaled steroids.
* Recent history of drug or alcohol abuse.
* Positive stool test for bacterial pathogens, Clostridium difficile toxin, or ovum and parasites.
* Vaccination within 28 days prior to randomization.
* Allergies to budesonide or to any other items used in its preparation.
* Participation in another clinical trial in the past 30 days.
* Pregnant or at risk of pregnancy.
* Taking a prohibited medication. Some medications to treat UP/UPS are prohibited during participation in the study, including laxatives and anti-diarrhea medications; however, oral 5-ASA agents at doses up to 4.8 g/day and daily fiber supplements are allowed. Other medications (e.g., antibiotics, anti-seizure and anti-coagulant medicines) are also prohibited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2009-11-17 (Actual); Primary Completion 2013-04-29 (Actual); Study Completion 2013-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director — Bausch Health Companies
Locations (63):
- United States (63):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Jonesboro, Arkansas
  - National City, California
  - Oakland, California
  - Orange, California
  - San Carlos, California
  - San Diego, California
  - Lakewood, Colorado
  - Littleton, Colorado
  - Bridgeport, Connecticut
  - Boynton Beach, Florida
  - Hollywood, Florida
  - Inverness, Florida
  - Largo, Florida
  - Maitland, Florida
  - Miami, Florida
  - New Smyrna Beach, Florida
  - Port Orange, Florida
  - Tampa, Florida
  - Trinity, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Newnan, Georgia
  - Bolingbrook, Illinois
  - Clive, Iowa
  - Baton Rouge, Louisiana
  - Shreveport, Louisiana
  - Lutherville, Maryland
  - Weymouth, Massachusetts
  - Troy, Michigan
  - Wyoming, Michigan
  - Jackson, Mississippi
  - Mexico, Missouri
  - St Louis, Missouri
  - Elizabeth, New Jersey
  - Vineland, New Jersey
  - Lake Success, New York
  - Boone, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Huntersville, North Carolina
  - LaPorte, North Carolina
  - Morganton, North Carolina
  - Cincinnati, Ohio
  - Gallipolis, Ohio
  - Mentor, Ohio
  - Norman, Oklahoma
  - Pittsburgh, Pennsylvania
  - Columbia, South Carolina
  - Franklin, Tennessee
  - Germantown, Tennessee
  - Jackson, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Bellevue, Washington
  - Vancouver, Washington
  - Milwaukee, Wisconsin

REFERENCES:
- [Derived] Bosworth BP, Sandborn WJ, Rubin DT, Harper JR. Baseline Oral 5-ASA Use and Efficacy and Safety of Budesonide Foam in Patients with Ulcerative Proctitis and Ulcerative Proctosigmoiditis: Analysis of 2 Phase 3 Studies. Inflamm Bowel Dis. 2016 Aug;22(8):1881-6. doi: 10.1097/MIB.0000000000000860. PMID 27416045
- [Derived] Sandborn WJ, Bosworth B, Zakko S, Gordon GL, Clemmons DR, Golden PL, Rolleri RL, Yu J, Barrett AC, Bortey E, Paterson C, Forbes WP. Budesonide foam induces remission in patients with mild to moderate ulcerative proctitis and ulcerative proctosigmoiditis. Gastroenterology. 2015 Apr;148(4):740-750.e2. doi: 10.1053/j.gastro.2015.01.037. Epub 2015 Jan 30. PMID 25644096

RESULTS

PARTICIPANT FLOW:
Groups:
- Budesonide: Participants who were diagnosed with active mild to moderate ulcerative proctitis (UP) or ulcerative proctosigmoiditis (UPS), received 2 milligrams (mg)/25 milliliter (mL) of budesonide foam, rectally twice daily for a period of 2 weeks followed by 2 mg/25 mL of budesonide foam, rectally once daily for a period of 4 weeks.
- Placebo: Participants who were diagnosed with active mild to moderate UP or UPS received 25 mL of placebo matching to budesonide foam twice daily for a period of 2 weeks followed by once daily for a period of 4 weeks.
Period: Overall Study
Arm/Group | Budesonide | Placebo
Started | 133 | 132
Received at Least 1 Dose of Study Drug | 133 | 132
Completed | 108 | 116
Not Completed | 25 | 16
Not completed — Adverse Event | 13 | 7
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Noncompliance | 1 | 0
Not completed — Low Cortisol | 2 | 0
Not completed — Lack of Efficacy | 2 | 6
Not completed — Met Exclusion Criterion | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Budesonide: Participants who were diagnosed with active mild to moderate (UP or UPS, received 2 mg/25 mL of budesonide foam, rectally twice daily for a period of 2 weeks followed by 2 mg/25 mL of budesonide foam, rectally once daily for a period of 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Budesonide | Placebo | Total
Number analyzed (Participants) | 133 | 132 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (13.94) | 41.4 (13.24) | 42.4 (13.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 80 | 152
  Male | 61 | 52 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 22 | 42
  Not Hispanic or Latino | 113 | 110 | 223
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 5 | 20
  White | 115 | 123 | 238
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Remission
Description: Remission was a combined assessment of clinical and endoscopic variables, defined as an endoscopy score of less than or equal to (<=) 1, a rectal bleeding score of 0, and an improvement or no change from baseline in stool frequency subscales of the Modified Mayo Disease Activity Index (MMDAI) at the end of 6 weeks of treatment. MMDAI was used to assess the overall disease activity for each participant. MMDAI evaluated 4 indices: stool frequency, rectal bleeding, physician's global assessment (PGA) and endoscopy findings each on a scale of 0 to 3 with a maximum total score of 12. Stool frequency MMDAI subscore ranged from 0-3, where 0 indicated normal number of stools per day and 3 indicated 5 or more stools than normal. Rectal bleeding MMDAI subscore ranged from 0-3, where 0 indicated no blood seen and 3 indicated blood alone passed. Endoscopy MMDAI subscore ranged from 0-3, where 0 indicated normal or inactive disease and 3 indicated severe disease (spontaneous bleeding, ulceration).
Time Frame: Week 6
Population: ITT population included all randomized participants. Missing data was imputed using last observation carried forward (LOCF) method.
Measure: Number; unit: percentage of participants
Groups:
- Budesonide: Participants who were diagnosed with active mild to moderate UP or UPS, received 2 mg/25 mL of budesonide foam, rectally twice daily for a period of 2 weeks followed by 2 mg/25 mL of budesonide foam, rectally once daily for a period of 4 weeks.
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 133 | 132
percentage of participants | 38.3 | 25.8
Statistical Analysis 1: Comparison: Budesonide vs Placebo; The logistic regression test was used to test for a difference in the percentages between the 2 treatment arms after adjusting for analysis center (country); Test type: Superiority; p = 0.0324, Regression, Logistic — Threshold for significance at 0.05 level

2. Secondary Outcome: Percentage of Participants Who Achieved a Rectal Bleeding MMDAI Subscale Score of 0 at End of Week 6
Description: The MMDAI was used to assess the overall disease activity for each participant. The MMDAI evaluated 4 indices:stool frequency, rectal bleeding, physician's global assessment and endoscopy findings each on a scale of 0 to 3 with a maximum total score of 12. Rectal bleeding MMDAI subscore ranged from 0-3, where 0 indicated no blood seen and 3 indicated blood alone passed. Missing data was imputed using LOCF method.
Time Frame: Week 6
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 133 | 132
percentage of participants | 46.6 | 28.0

3. Secondary Outcome: Number of Scheduled Assessments With Rectal Bleeding Responder Classification
Description: The MMDAI was used to assess the overall disease activity for each participant. The MMDAI evaluated 4 indices: stool frequency, rectal bleeding, physician's global assessment and endoscopy findings each on a scale of 0 to 3 with a maximum total score of 12. Rectal bleeding MMDAI subscore ranged from 0-3, where 0 indicated no blood seen and 3 indicated blood alone passed. Percentage of participants who were rectal bleeding responder at scheduled assessments were reported. Rectal bleeding responders were defined as those participants who achieved a rectal bleeding MMDAI subscale score of 0 during the treatment period. Missing data was imputed using LOCF method.
Time Frame: Weeks 1, 2, 4, and 6
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 133 | 132
percentage of participants
  Responder at 1 Assessment | 12.0 | 13.6
  Responder at 2 Assessment | 18.8 | 13.6
  Responder at 3 Assessment | 21.1 | 10.6
  Responder at 4 Assessment | 6.0 | 1.5

4. Secondary Outcome: Percentage of Participants Who Achieved an Endoscopy MMDAI Subscale Score of 0 or 1 at End of Week 6
Description: The MMDAI was used to assess the overall disease activity for each participant. The MMDAI evaluated 4 indices: stool frequency, rectal bleeding, physician's global assessment and endoscopy findings each on a scale of 0 to 3 with a maximum total score of 12. Endoscopy subscale ranged from 0-3, where 0 = normal or inactive disease, 1 = mild disease, 2 = moderate disease and 3 = severe disease (spontaneous bleeding, ulceration). Percentage of participants with normal or mild disease have been presented in this outcome measure. Missing data was imputed using LOCF method.
Time Frame: Week 6
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 133 | 132
percentage of participants | 55.6 | 43.2

5. Secondary Outcome: Percentage of Participants Who Achieved a Score of 0 for Rectal Bleeding Subscale and a Combined Score of <=2 for Bowel Frequency and Physician's Global Assessment (PGA) in the MMDAI Subscales at End of Week 6
Description: The MMDAI was used to assess the overall disease activity for each participant. The MMDAI evaluated 4 indices: stool frequency, rectal bleeding, PGA and endoscopy findings each on a scale of 0 to 3 with a maximum total score of 12. Rectal bleeding subscore ranged from 0-3, where 0 indicated no blood seen and 3 indicated blood alone passed. Bowel frequency (BF) subscore ranged from 0-3, where 0 indicated normal number of stools per day and 3 indicated 5 or more stools than normal. PGA subscore ranged from 0-3, where 0 indicated normal disease and 3 indicated severe disease. Missing data was imputed using LOCF method.
Time Frame: Week 6
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 133 | 132
percentage of participants | 41.4 | 25.8

6. Secondary Outcome: Percentage of Participants Who Achieved an MMDAI Total Score of <= 3 With Greater Than or Equal to (>=2) Points of Improvement From Baseline at the End of Week 6
Description: The MMDAI was used to assess the overall disease activity for each participant. The MMDAI evaluated 4 indices: stool frequency, rectal bleeding, physician's global assessment and endoscopy findings each on a scale of 0 to 3 with a maximum total score of 12. Rectal bleeding subscore ranged from 0-3, where 0 indicated no blood seen and 3 indicated blood alone passed. BF subscore ranged from 0-3, where 0 indicated normal number of stools per day and 3 indicated 5 or more stools than normal. Physician global assessment (PGA) subscore ranged from 0-3, where 0 indicated normal and 3 indicated severe disease. Endoscopy subscore ranged from 0-3, where 0 indicated normal and 3 indicated severe disease. MMDAI total score ranged from 0-12, where higher score indicated severe disease. Missing data was imputed using LOCF method.
Time Frame: Week 6
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 133 | 132
percentage of participants | 45.9 | 30.3

7. Secondary Outcome: Percentage of Participants Who Achieved Improvement of >=1 Point From Baseline in the MMDAI Endoscopy Subscale Score at End of Week 6
Description: The MMDAI was used to assess the overall disease activity for each participant. The MMDAI evaluated 4 indices: stool frequency, rectal bleeding, PGA and endoscopy findings each on a scale of 0 to 3 with a maximum total score of 12. Endoscopy subscore ranged from 0-3, where 0 = normal or inactive disease, 1 = mild disease (erythema, decreased vascular pattern), 2 = moderate disease (marked erythema, absent vascular pattern, friability, erosions), and 3 = severe disease (spontaneous bleeding, ulceration). Missing data was imputed using LOCF method.
Time Frame: Week 6
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 133 | 132
percentage of participants | 57.1 | 47.7

8. Secondary Outcome: Percentage of Participants Who Achieved Improvement of >=1 Point From Baseline in the MMDAI Rectal Bleeding Subscale Score at End of Week 6
Description: The MMDAI was used to assess the overall disease activity for each participant. The MMDAI evaluated 4 indices: stool frequency, rectal bleeding, PGA and endoscopy findings each on a scale of 0 to 3 with a maximum total score of 12. Rectal bleeding MMDAI subscore ranged from 0-3, where 0 = no blood seen, 1 = streaks of blood with stool less than half the time, 2 = obvious blood with stool most of the time, and 3 indicated blood alone passed. Missing data was imputed using LOCF method.
Time Frame: Week 6
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 133 | 132
percentage of participants | 70.7 | 53.0

9. Secondary Outcome: Percentage of Participants Who Achieved >=3 Point Improvement From Baseline in the MMDAI Total Score Including Improvement of >=1 Point From Baseline in the MMDAI Rectal Bleeding Subscale Score and MMDAI Endoscopy Subscale at End of Week 6
Description: The MMDAI was used to assess the overall disease activity for each participant. The MMDAI evaluated 4 indices: stool frequency, rectal bleeding, PGA and endoscopy findings each on a scale of 0 to 3 with a maximum total score of 12. Rectal bleeding subscore ranged from 0-3, where 0 indicated no blood seen and 3 indicated blood alone passed. BF subscore ranged from 0-3, where 0 indicated normal number of stools per day and 3 indicated 5 or more stools than normal. PGA subscore ranged from 0-3, where 0 indicated normal and 3 indicated severe disease. Endoscopy subscore ranged from 0-3, where 0 indicated normal and 3 indicated severe disease. MMDAI total score ranged from 0-12, where higher score indicated severe disease. Missing data was imputed using LOCF method.
Time Frame: Week 6
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 133 | 132
percentage of participants | 52.6 | 37.9

10. Secondary Outcome: Mean Change From Baseline to Week 6 in MMDAI Total Score and Subscale Scores
Description: as for outcome 9
Time Frame: Baseline, Week 6
Population: ITT population included all randomized participants.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 133 | 132
unit on a scale
  Bowel frequency score: Baseline | 1.8 (0.87) | 1.9 (0.93)
  Bowel frequency score: Change at Week 6 | -0.7 (0.98) | -0.5 (0.85)
  Rectal Bleeding score:Baseline | 2.1 (0.38) | 2.1 (0.36)
  Rectal Bleeding score: Change at Week 6 | -1.2 (0.95) | -0.8 (0.93)
  PGA score:Baseline | 1.8 (0.43) | 1.8 (0.41)
  PGA score: Change at Week 6 | -0.8 (0.79) | -0.5 (0.78)
  Endoscopy score:Baseline | 2.1 (0.30) | 2.1 (0.29)
  Endoscopy score: Change at Week 6 | -0.8 (0.76) | -0.5 (0.74)
  Total score:Baseline | 7.8 (1.23) | 7.9 (1.28)
  Total score: Change at Week 6 | -3.5 (2.80) | -2.4 (2.74)

ADVERSE EVENTS:
Time Frame: From start of study drug up to Week 8
Description: Safety population included all randomized participants who were administered at least one dose of the study drug. 1 participant was randomized to placebo, but received both placebo and budesonide during study. This participant was analyzed in placebo group in all efficacy analyses and is summarized in budesonide group in all safety analyses.
Arm/Group | Budesonide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/134 | 0/131
Serious Adverse Events (participants affected / at risk) | 2/134 | 3/131
Other Adverse Events (participants affected / at risk) | 66/134 | 47/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Budesonide (N=134) | Placebo (N=131)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/72 | 1/80 — This is a gender-specific AE. Only female participants were at risk.
Arterial thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Budesonide (N=134) | Placebo (N=131)
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Proctitis ulcerative (Gastrointestinal disorders) | 0 | 4
Blood bilirubin increased (Investigations) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Tongue geographic (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Acute sinusitis (Infections and infestations) | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2
Colitis ulcerative (Gastrointestinal disorders) | 1 | 2
Oedema peripheral (General disorders) | 0 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Nipple pain (Reproductive system and breast disorders) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Abdominal tenderness (Gastrointestinal disorders) | 1 | 2
Proctalgia (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 4 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Rectal prolapse (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Anal pruritus (Gastrointestinal disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Acute tonsillitis (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Application site pain (General disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Eye swelling (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 0 | 1
Blood cortisol decreased (Investigations) | 25 | 0
Blood glucose abnormal (Investigations) | 1 | 0
ACTH stimulation test abnormal (Investigations) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 7 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Purpura senile (Skin and subcutaneous tissue disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2
Headache (Nervous system disorders) | 4 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/72 | 0/80 — This is a gender-specific AE. Only female participants were at risk.
Sexual dysfunction (Reproductive system and breast disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.